CLINICAL TRIAL: NCT03268252
Title: Optimization of Mass Drug Administration With Existing Drug Regimens for Lymphatic Filariasis: Monitoring Efficacy of Ongoing Treatment Programs in Papua New Guinea
Brief Title: Optimization of MDA With Existing Drug Regimens for LF: Monitoring Efficacy of Ongoing Treatment Programs in PNG
Acronym: MDA
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government)
Responsible Party: Principal Investigator, Christopher L. King, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: CWRU Optimization MDA LF PNG
Record Dates: First submitted 2013-10-28; First posted 2017-08-31 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Lymphatic Filariasis
MeSH Terms: conditions — Elephantiasis, Filarial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any remaining from the finger stick/stool samples will be cryopreserved for subsequent testing for presence of other infections that have public health importance in PNG (e.g., malaria) using molecular or serological assays. Genetic testing of samples for the LF, malaria or common blood borne or intestinal infections will be performed using microsatellite markers or highly polymorphic genes as confirmatory diagnostic tests and/or to assess the diversity of the parasite populations in the communities.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2x/year MDA: Diethylcarbamazine 6 mg/kg + Albendazole 400 mg given twice per year
- 1x/year MDA: Diethylcarbamazine 6 mg/kg + Albendazole 400 mg given once per year

SUMMARY:
The standard regimen for elimination of lymphatic filariasis (LF) in PNG is annual administration of two drugs at the same time. The two drugs are called "DEC" (Diethylcarbamazine, 6 mg/kg body weight) and "ALB" (Albendazole 400 mg for all individuals regardless of weight), which are given one time per year for five to seven years with the aim to interrupt transmission that occurs through local mosquito vectors. These drugs kill the larval forms of the parasite in the blood that are necessary for continuing transmission of infection by the mosquito vector. The two drugs were previously thought to have little effect on adult worms, the stage of the parasite which is responsible for production of the larval forms that appear in the blood of infected people. Recent data, however, suggest that DEC and ALB can kill or render adult worms unable to produce the larval forms (sterilization). Therefore, giving these drugs twice per year for three consecutive years may increase the rate of killing or sterilizing of adults worms over regimens that involve administration of the same drugs only one time per year. The overall goal of this research is to compare the anti-parasite activity of DEC plus ALB given one time per year, the current standard for MDA to eliminate LF, to DEC plus ALB given two times per year (at 6-month intervals) in order to reduce the total duration and cost of MDA to eliminate LF in PNG. Adults (18 years and older) and minors (age 5 to 17 years) will be invited to participate in this study. Study participants will be asked to give finger stick blood samples to check LF infection status and stool samples to determine how well the drugs eliminate intestinal worm infections. Sampling will be done by repeated cross-sectional surveys in the same communities, but not necessarily the same persons, one time per year over a 3-year period. As part of the annual treatment infection surveillance the study team will also collect demographic data (place of residence, family relationship, age, use of bed nets), history of swelling of the arms and legs (elephantiasis), scrotal swelling (hydrocele), acute filarial fever accompanied by extremity swelling, and history of prior treatment for LF.

DETAILED DESCRIPTION:
This research will conduct a population-based field studies to determine whether the relative cost and efficacy of semi-annual versus annual administration of MDA using DEC (6 mg/kg body weight) plus ALB 400 mg (for all individuals regardless of weight) will be more successful in elimination of LF and reduction in the burden of soil transmitted helminth (worm) infections. The study involving participation of human subjects is observational in nature, uses drugs that are the standard approved treatment for LF in PNG and elsewhere in the Pacific and Asia, and does not involve administration of drugs by the investigators. Diagnosis of LF and administration of anti-LF drugs will be the responsibility of those authorized by the PNG Department of Health to perform this activity.

The study design is repeated cross-sectional surveys examining each subject once. Some subjects may be included in more than one annual population survey, but this is not a longitudinal study. Approximately 3,200 individuals will participate per year at the beginning of the study and at years 1, 2 and 3 (a total of 4 cross-sectional surveys). The study will include both females and males 5 years of age and older who live in a LF endemic area of PNG. Subject selection will not be based on health status. The study aims to determine the relative impact and cost effectiveness of annual versus twice yearly MDA (DEC 6 mg/kg body plus Alb 400 mg for all individuals) for elimination of LF and reduction in soil transmitted helminthic infection burdens in these populations.

The project is comprised of repeated annual cross-sectional surveys in sentinel communities before and after initiation of MDA for LF. The surveys will be conducted over a period of 3 years at the following times: 0 (pre-treatment baseline), 1, 2, and 3 years corresponding to annual treatment times. Government health officials as part of the GPELF will administer the MDA (standard regimen recommended by WHO is DEC + ALB). Part of the government-sponsored program will be to screen for LF using ICT card screening and finger stick bloods for measuring the density of blood born microfilaria (MF). The current protocol will assist in collection of these data. As part of the annual treatment infection surveillance the study team will also collect demographic data, history of lymphedema, scrotal swelling (hydrocele), acute filarial fever or adenolymphangitis, and history of prior treatment for LF.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged >=5 years of age in the community
2. Willingness to give informed consent to participate in the study
3. Willingness of parents or guardians to give consent for minors to participate in study

Exclusion Criteria:

1. Not willing or able to give informed consent for the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population (3,200/survey) will include male and female subjects >=5 years of age living in East Sepik Province, PNG. If unexpected logistical problems should arise, other study areas have been identified in Madang Province. The proposed study area will be in the Dreikikier Rural Local Level Government (LLG, approx pop 20,000) and Gawanga Rural, LLG (approx pop 13,000). Residents of villages previously treated with MDA will not be included in the study.
  Children <5 years of age from community studies excluded because prevalence rates for LF tend to be very low in young children and because of difficulties associated with collecting clinical specimens from this population. Pregnancy will not be an exclusion criteria because DEC and ALB are considered safe in pregnancy.
Sampling Method: Probability Sample
Enrollment: 3200 (Actual)
Dates: Start 2012-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The comparator (standard treatment) DEC 6mg/kg + Alb 400mg administered annually (at 0, 12 and 24 months). | 36 months
  Determine if administering DEC 6 mg/kg + ALB 400 mg given twice per year is more effective than standard DEC 6 mg/kg + Alb 400 mg given once per year in achieving reduction of microfilarial prevalence caused by Wuchereria bancrofti infection to less than 1% at 36 months after the initiation of the study.

SECONDARY OUTCOMES:
DEC 6mg/kg + Alb 400 given once | 36 months
  We will test the hypothesis that twice annual MDA is superior to annual MDA for achieving a significantly greater reduction in prevalence and intensity of infection of STH infection infections at 36 months after the initiation of the study
DEC 6 mg/kg + Alb 400 mg + Iver 200 µg/kg administered once only at the beginning of the RCT (0 month). | 36 months
  We will test the hypothesis that twice annual MDA is more cost effective compared to annual MDA for eliminating LF at 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: James W Kazura, MD, Principal Investigator — Case Western Reserve University; Christopher L King, MD, PhD, Principal Investigator — Case Western Reserve University; Peter M Siba, PhD, Principal Investigator — Papua New Guinea Institute of Medical Research
Locations (1):
- Papua New Guinean Institute for Medical Research, Maprik, Sandaun Province, Papua New Guinea